CLINICAL TRIAL: NCT01326156
Title: Patellofemoral Arthroplasty (PFA) Versus Total Knee Replacement (TKR) for Isolated Patellofemoral Osteoarthritis
Brief Title: Study of Knee Replacements for Patellofemoral Osteoarthritis
Acronym: PFA/TKR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Stryker Nordic (Industry); DePuy Orthopaedics (Industry); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56789
Record Dates: First submitted 2009-05-19; First posted 2011-03-30 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis, Knee; Patellofemoral Knee Arthroplasty
Keywords: Osteoarthritis; Knee; Knee cap; Patella; Patellofemoral
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Patella Fracture | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Pragmatic, multi-centre, 1:1 parallel-group, randomised controlled trial. Double-blinded for 1st year. PROMs completion without staff involvement. Statistical consultants blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients are blinded to treatment allocation for the first year; they are un-blinded at the one-year follow-up. Hospital staff, excluding the surgical team, are likewise blinded. Discharge letters are intended to exclude implant information to ensure general practitioner blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avon patellofemoral replacement (Experimental): Knee arthroplasty with insertion of patellofemoral joint replacement.
  Interventions: Device: Knee arthroplasty
- PFC Sigma CR total knee replacement (Active Comparator): Knee arthroplasty with total (tricompartmental) knee replacement.
  Interventions: Device: Knee arthroplasty

INTERVENTIONS:
Device: Knee arthroplasty — Comparison of patellofemoral arthroplasty versus conventional total knee arthroplasty in cases of isolated patellofemoral osteoarthritis.
  Other Names: PFA: Avon Patellofemoal arthroplasty (Stryker); TKR: PFC Sigma CR arthroplasty (DePuy)

SUMMARY:
This is a randomized comparison of PFA and TKR in treatment of isolated patellofemoral osteoarthritis.

DETAILED DESCRIPTION:
Isolated patellofemoral osteoarthritis can be a disabling condition of the knee necessitating knee arthroplasty. It is debated whether total knee replacement or isolated patellofemoral replacement is the better treatment option. This randomized trial attempts to give a qualified answer to the debate by comparing clinical outcome (range of movement, stability, effusion, patellofemoral tracking, tenderness, stair climbing), patient self assessment scores (EQ-5D, Oxford Knee Score, KOOS, SF-36, AKS), complications (infections, revisions), longevity (survival analysis) and cost (direct and indirect) for the two implant types.

The Avon patellofemoral implant has been chosen, as this is the patellofemoral implant with the best documentation. The PFC Sigma CR total knee implant has been chosen as it a current standard implant and market leader.

ELIGIBILITY:
Inclusion Criteria:

* Isolated PF-OA

Exclusion Criteria:

* Medial or lateral OA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2025-04 (Actual); Study Completion 2040-10 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcomes (disease-specific and generic QoL instruments) | 10 years
  The physical functioning score of the Short Form (36) Health Survey is the primary outcome measure of the study. Disease-specific patient-reported outcomes (Oxford Knee Score, KOOS and Kujala) and a second generic quality of life measure (EQ5D).

SECONDARY OUTCOMES:
Implant survival, clinician assessment and cost. | 10 years
  Secondary outcome measures relate to implant survival, clinician assessment and cost. Implant survival will be assessed by 5- and 10-year implant survival rates and by analyzing causes for revision surgery. Clinician assessment includes Knee Society Score (stability, range of movement, effusion, tenderness etc.). Assessments of immediate and long-term costs are based on patient diaries, sick leave, use of medical services and drug prescriptions.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Odgaard, FRCS, DMSc, Principal Investigator — Dept. of Orthopaedics, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in published article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 6 months and and ending 5 years following article publication.
Access Criteria: For investigators whose proposed use of the data has been approved by and independent review committee identified for this purpose or for researchers who provide a methdologically sound proposal.
  Types of analyses accepted: For acheiving aims of the approved proposal.
  Proposals should be directed to anders.odgaard@regionh.dk. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years following publication at a third party website.

REFERENCES:
- [Result] Martinique VB, Julie H, Snorre S, Soeren R, Kristensen WP, Zahid A, Alex L, Justin C, Anders O. Equivocal Physical Activity Outcomes 10 Years After Patellofemoral vs Total Knee Replacement: Follow-Up of a Previously Reported Randomised Controlled Trial in Isolated Patellofemoral Joint Osteoarthritis. J ISAKOS. 2025 Nov 15:101037. doi: 10.1016/j.jisako.2025.101037. Online ahead of print. PMID 41248881
- [Result] Odgaard A, Kappel A, Madsen F, Kristensen PW, Stephensen S, Attarzadeh AP. Erratum to: Patellofemoral Arthroplasty Results in Better Time-weighted Patient-reported Outcomes After 6 Years than TKA: A Randomized Controlled Trial. Clin Orthop Relat Res. 2023 Jul 1;481(7):1455-1457. doi: 10.1097/CORR.0000000000002713. Epub 2023 Jun 15. No abstract available. PMID 37352486
- [Result] Odgaard A, Kappel A, Madsen F, Kristensen PW, Stephensen S, Attarzadeh AP. Patellofemoral Arthroplasty Results in Better Time-weighted Patient-reported Outcomes After 6 Years than TKA: A Randomized Controlled Trial. Clin Orthop Relat Res. 2022 Sep 1;480(9):1707-1718. doi: 10.1097/CORR.0000000000002178. Epub 2022 Mar 21. PMID 35315804
- [Result] Fredborg C, Odgaard A, Sorensen J. Patellofemoral arthroplasty is cheaper and more effective in the short term than total knee arthroplasty for isolated patellofemoral osteoarthritis: cost-effectiveness analysis based on a randomized trial. Bone Joint J. 2020 Apr;102-B(4):449-457. doi: 10.1302/0301-620X.102B4.BJJ-2018-1580.R3. PMID 32228074
- [Result] Odgaard A, Madsen F, Kristensen PW, Kappel A, Fabrin J. The Mark Coventry Award: Patellofemoral Arthroplasty Results in Better Range of Movement and Early Patient-reported Outcomes Than TKA. Clin Orthop Relat Res. 2018 Jan;476(1):87-100. doi: 10.1007/s11999.0000000000000017. PMID 29529622